CLINICAL TRIAL: NCT06143384
Title: Benefits of Telemonitoring in Home Mechanical Ventilation by the Use of a Simple and Intuitive Algorithm
Brief Title: Telemonitoring in Home Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erasme University Hospital (Other)
Collaborators: Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Michel Toussaint, Coordinator Center for Home Mechanical Ventilation, Erasme University Hospital
Other Study IDs: Citadelle Liège project1
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Insufficiency Requiring Mechanical Ventilation
Keywords: home mechanical ventilation; telemonitoring

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients using Home Mechanical Ventilation (HMV): Patients using Home Mechanical Ventilation (HMV), and registered in the Belgian agreement for HMV at 1/ the Citadelle hospital in Liège, Belgium and 2/HUB-Erasme hospital, Brussels, Belgium.
  Interventions: Device: Telemonitoring AirView (ResMed company)

INTERVENTIONS:
Device: Telemonitoring AirView (ResMed company) — Introduction of AirView telemonitoring of HMV, during a 6-months period.

SUMMARY:
Multicentric, observational and longitudinal prospective evaluation of build-in-software data telemonitoring of home ventilators in patients using Home Mechanical Ventilation in Belgium.

DETAILED DESCRIPTION:
OBJECTIVES : Use of a decisional algorithm (developed by La Citadelle/Liège) to assess Telemonitoring (AirView type, ResMed) of data in the ventilators of patients using Home Mechanical Ventilation (HMV), and registered in the Belgian agreement for HMV at 1/ the Citadelle hospital in Liège and 2/HUB-Erasme, Brussels, Belgium.

BACKGROUND: HMV initiated in the hospital is used at home. Patients who benefit from HMV present significant functional limitations of cardio-respiratory, neurological and/or physical origin. Such limitations compromise the ability of patients to travel to the referring hospital. As a result, good treatment follow-up is difficult to assess both from quantity and quality points of view. This is why Telemonitoring systems have been developed to access ventilator build-in-software data at through dedicated online systems. In other words, data from devices operating at home can be sent to the hospital and analyzed in real time by professionnals in the hospital. This project aims to evaluate the impact of Telemonitoring ventilator's data on the quality of HMV-monitoring in patients living and using HMV at home.

METHODS: A one-year multicentric, observational, longitudinal and prospective evaluation of build-in-software data telemonitoring of home ventilators in patients using HMV in Belgium. The two Belgian hospitals will each follow 10 patients for one year (2024). The data from the ventilator as well as the actions to be taken in response to Airview Telemonitoring alerts will be carried out using a decision-making algorithm created by the Citadelle Hospital in Liège.

ELIGIBILITY:
Inclusion Criteria:

* All patients starting HMV in 2024, followed up in 1/ Liège or 2/ Brussels, and using devices from the ResMed company (Astral 150 ou Lumis 150).

Exclusion Criteria:

* Individuals refusing to sign the consent form
* Presence of acute pathology requiring hospitalization and close monitoring of ventilation
* Patients using a tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring noninvasive ventilation at home and followed-up in Liège or Brussels hospitals, as previously described.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance to the treatment | T1: Mean value during night 1 (inpatient)
  Hours of use of HMV/24h
Compliance to the treatment | T2: Mean value during night 2 (inpatient)
  Hours of use of HMV/24h
Compliance to the treatment | T3: Mean value during nights 24-30 (outpatient)
  Hours of use of HMV/24h
Compliance to the treatment | T4: Mean value during nights 174-180 (outpatient)
  Hours of use of HMV/24h
Leaks | T1: Median value during night 1 (inpatient)
  Unintentional leaks inform about undesirable leakage around the mask (bad sealing) or patients mouth leakage.
Leaks | T2: Median value during nights 2 (inpatient)
  Unintentional leaks inform about undesirable leakage around the mask (bad sealing) or patients mouth leakage.
Leaks | T3: Median value during nights 24-30 (outpatient)
  Unintentional leaks inform about undesirable leakage around the mask (bad sealing) or patients mouth leakage.
Leaks | T4: Median value during nights 174-180 (outpatient)
  Unintentional leaks inform about undesirable leakage around the mask (bad sealing) or patients mouth leakage.
AHI index | T1 : Median value during night 1 (inpatient)
  The apnea-hypopnea index (AHI) informs about obstructive and apneic events during HMV.
AHI index | T2: Median value during night 2 (inpatient)
  The apnea-hypopnea index (AHI) informs about obstructive and apneic events during HMV.
AHI index | T3: Median value during nights 24-30 (outpatient)
  The apnea-hypopnea index (AHI) informs about obstructive and apneic events during HMV.
AHI index | T4: Median value during nights 174-180 (outpatient)
  The apnea-hypopnea index (AHI) informs about obstructive and apneic events during HMV.

SECONDARY OUTCOMES:
Inconfort score | T1 : Score after night 1 (inpatient)
  This score (0-4 points) evaluates the discomfort of the patient using HMV. A score of zero suggests perfect comfort (none out of the 4 symptoms present) and a score of 4 (all symptoms present) suggests maximal discomfort related to the presence of the following 4 symptoms: pain or skin lesions, dryness of the mucous membranes, rhinitis or eye irritation, discomfort related to the settings of the device.
Inconfort score | T2 : Score after night 2 (inpatient)
  This score (0-4 points) evaluates the discomfort of the patient using HMV. A score of zero suggests perfect comfort (none out of the 4 symptoms present) and a score of 4 (all symptoms present) suggests maximal discomfort related to the presence of the following 4 symptoms: pain or skin lesions, dryness of the mucous membranes, rhinitis or eye irritation, discomfort related to the settings of the device.
Inconfort score | T3 : Score after nights 24-30 (outpatient)
  This score (0-4 points) evaluates the discomfort of the patient using HMV. A score of zero suggests perfect comfort (none out of the 4 symptoms present) and a score of 4 (all symptoms present) suggests maximal discomfort related to the presence of the following 4 symptoms: pain or skin lesions, dryness of the mucous membranes, rhinitis or eye irritation, discomfort related to the settings of the device.
Inconfort score | T4 : Score after nights 174-180 (outpatient)
  This score (0-4 points) evaluates the discomfort of the patient using HMV. A score of zero suggests perfect comfort (none out of the 4 symptoms present) and a score of 4 (all symptoms present) suggests maximal discomfort related to the presence of the following 4 symptoms: pain or skin lesions, dryness of the mucous membranes, rhinitis or eye irritation, discomfort related to the settings of the device.
Algorithm Score | T2 : Score after night 2 (inpatient)
  This score (0-2 points) is given by the professional assessing the algorithm effectiveness after the Airview data analysis: 0 - no or useless intervention of the carer after using the algorithm, 1 - partial positive improvement after intervention post-algorithm, 2 - clear improvement after intervention post-algorithm or no use of the algorithm because of perfect use of HMV at home.
Algorithm Score | T3 : Score after nights 24-30 (outpatient)
  This score (0-2 points) is given by the professional assessing the algorithm effectiveness after the Airview data analysis: 0 - no or useless intervention of the carer after using the algorithm, 1 - partial positive improvement after intervention post-algorithm, 2 - clear improvement after intervention post-algorithm or no use of the algorithm because of perfect use of HMV at home.
Algorithm Score | T4 : Score after night 2 (outpatient)
  This score (0-2 points) is given by the professional assessing the algorithm effectiveness after the Airview data analysis: 0 - no or useless intervention of the carer after using the algorithm, 1 - partial positive improvement after intervention post-algorithm, 2 - clear improvement after intervention post-algorithm or no use of the algorithm because of perfect use of HMV at home.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy De Fooz, Dr, Study Director — Citadelle Hospital; Adrien Meunier, MSc, Principal Investigator — Citadelle Hospital
Locations (1):
- Michel Toussaint, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No